CLINICAL TRIAL: NCT03456622
Title: A Prospective, Observational, Multi-centre, Cohort Study of the G7™Acetabular System Used With Compatible Femoral Stems in Patients With Degenerative Disease of the Hip
Brief Title: BC Study of G7 Cup and Compatible Femoral Stems
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.GH59
Record Dates: First submitted 2018-01-12; First posted 2018-03-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non-inflammatory Degenerative Joint Disease; Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis
Keywords: G7
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective , observational, multi-centre, cohort study of the G7™ Acetabular System used with compatible femoral stems in patients with degenerative disease of the hip.

The study will be enrolled onto Beyond Compliance.

DETAILED DESCRIPTION:
The UK Beyond Compliance is a joint effort between implant manufacturers, implanting surgeons adopting our products, and the Beyond Compliance Advisory Group, all of whom are looking to ensure the safe and stepwise introduction of new or modified implants to the market in the interest of patients.

The G7 Acetabular Cup System is Biomet multi-bearing acetabular platform with a wide range of acetabular shell options recently launched. There is a need to provide evidence on the safety and performance of this cup to support the product in different markets.

The purpose of this multicenter study is to assess the clinical performance of the G7 acetabular system under standard condition of use. The data will help Biomet to gain 3A ODEP rating in 4 years and up to 10 year rating

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥18 years
* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis, suitable for unilateral primary hip replacement;
* Rheumatoid arthritis;
* Correction of functional deformity;
* Voluntary written Informed Consent obtained

Exclusion Criteria

Pre-operative:

* Prospect for recovery to independent mobility compromised by known coexistent medical problems;
* Requiring revision hip replacement;
* Requiring bilateral hip replacement;
* Previous hip replacement (resurfacing or THR) on the contralateral side and whose outcome is achieving an Oxford Hip score <18 points;
* Likely post-operative leg length inequality >5cm;
* Neuromuscular disease affecting hip (Parkinson's, cerebral palsy, other spasticity);
* Primary or metastatic tumour involving this hip;
* Loss of abductor musculature, poor bone stock, or poor skin coverage around the hip joint;
* Previous organ transplant;
* Previous arthrodesis or excision arthroplasty
* Abnormal acetabulum:

  * Acetabular deficiency - >2cm superior loss acetabular dome or >1.5cm protrusion acetabulae or wall deficiency> half a wall;
  * Dysplasia (DDH) with >2.5cm subluxation or complete dislocation;
* Body mass index > 40kg/m2;
* Active or previous or suspected infection in this hip;
* Sepsis or osteomyelitis;
* Known sensitivity to device materials;
* Women judged by the investigator to be of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period;
* Unable to provide informed consent (insufficient English, cognitive disorder such as dementia, psychiatric illness);
* Unable to complete follow-ups (life expectancy <5 years, insufficient English, lives overseas, unable to return easily).

Intra-operative:

* Abnormal abductor mechanism - trochanter escape > 1.5cm or gluteus medius totally non-functional or trochanter absence;
* Unavailability of required size of prosthesis;
* Abnormal acetabulum:

  * Acetabular deficiency - >2cm superior loss acetabular dome or >1.5cm protrusion acetabulae or wall deficiency> half a wall;
  * Dysplasia (DDH) with >2.5cm subluxation or complete dislocation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals who receive the study device, meet inclusion/exclusion criteria and provided nformed consent.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival of the implant system | 10 years post-surgery
  Survival of the implant based on removal or intended removal of any component

SECONDARY OUTCOMES:
Oxford Hip Score | pre-op, 6 Months, 1 Year, 3 Year
  The Oxford Hip Score (OHS) is a patient-reported outcome measure that was developed to specifically assess the patient's perspective of outcome following THA. The OHS consists of twelve questions covering function and pain associated with the hip. To calculate the total score, each response is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27
Harris Hip Score | pre-op, 1 Year, 3 Year
  The Harris Hip Score (HHS) is an outcome measure that includes a series ofquestions answered by the patient and physical examinations recorded by aqualified health care professional. The HHS covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence ofdeformity (one item, 0-4 points) and range of motion (one item, 0-5 points). Toobtain a final score, the points are summed. The outcome score can be categorizedas Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70
EQ-5D-3L score | pre-op, 6 Months, 1 Year, 3 Year
  The EQ-5D-3L is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes five dimensions referring to mobility, self-care, daily activities,pain/discomfort, and anxiety/depression. Each question can be answered in three ways/levels indicating no problems, some problems, and extreme problems. In the derived EQ-5D-3L score, the highest score is 1 and the lowest score is -0.594; negative numbers correspond to a self-assessed health state worse than being dead.
EQ-5D-3L VAS | pre-op, 6 Months, 1 Year, 3 Year
  The EQ-5D-3L is a standardized instrument widely used to measure health status.It is a self-reported assessment about the patient's quality of life. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The VAS is a vertical scale ranging from 100 ('The best health you can imagine') to 0 ('The worst health you can imagine') where the patient reports his/her current state of health.
Hip disability and Osteoarthiritis Outcome Score (HOOS) | pre-op, 6 Months, 1 Year, 3 Year
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a questionnaire designed to assess patient-relevant outcomes of hip related problems [Nilsdotter et al., 2003]. The HOOS covers five domains: pain (ten items), symptoms (five items), activity of daily living (17 items), sport/recreation function (four items), and hip-related quality of life (QoL) (four items). All items have five possible answer options scored from 0 (no problems) to 4 (extreme problems). The mean scores of each domain are transformed to a 0-100 scale, with 0 representing extreme hip problems and 100 representing no hip problems.
Radiographic assessment | 1 year post-op
  Assessing radiolucency
Radiographic assessment | post-op, 2-8 weeks, 1 Year, 3 Year
  Assessing radiolucency
Safety of the implant system | 10 years post-surgery
  Safety of the system will be assessed by monitoring the frequency and incidence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Bournemouth Hospital, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No